CLINICAL TRIAL: NCT01853956
Title: Open,Two-period, Two-treatment, Two-sequence, Cross-over, Randomized Trial of Single Doses of Two Oral Preparations With 0.25 mg of Alprazolam (Zamoprax® GlaxoSmithKline México, S.A. de C.V. vs. Tafil® 0.25mg, Pharmacia &Upjohn, S.A. de C.V.) in Fasting Healthy Volunteers
Brief Title: Bioequivalence Trial of Alprazolam 0.25 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116937
Record Dates: First submitted 2012-11-28; First posted 2013-05-15 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Anxiety Disorders
Keywords: Mexico; Bioequivalence; Alprazolam; Pharmacokinetics
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (reference)/ B (test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Alprazolam 0.25 mg
- B (test)/ A (reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Alprazolam 0.25 mg

INTERVENTIONS:
Drug: Alprazolam 0.25 mg — Reference product
  Other Names: Tafil®; Pharmacia & Upjohn
Drug: Alprazolam 0.25 mg — Test product
  Other Names: Zamoprax®; GlaxoSmithKline

SUMMARY:
The objective of this study was to confirm if two formulations of alprazolam (tablets) are bioequivalent.

Test product was Zamoprax® 0.25 mg (GlaxoSmithKline) and reference product Tafil® 0.25 mg (Pharmacia & Upjohn). One tablet was the single dosage.

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fasting conditions.

The population was composed of 28 healthy volunteers, both genders, adults between 18-50 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

* Free will participation according to Mexican regulation, Helsinki Declaration, and Good Clinical Practice.
* Healthy, between 18 and 50 years.
* Body Mass Index between 18 and 27.5
* In good health by complete medical history and laboratory tests.
* Blood pressure 130-90/ 90-60 mm Hg; heart rate 55-100 beat per minute, respiratory rate 14-20 movements per minute.
* Laboratory tests +/- 10% of normal interval (blood cytology, blood chemistry 27 elements, Hepatitis B and C antigens, HIV, urinalysis, anti-doping, pregnancy, electrocardiogram

Exclusion Criteria:

* Alteration of vital signs
* Not complying with inclusion criteria
* History of cardiovascular, kidney, hepatic, muscular, metabolic, gastrointestinal (including constipation), neurologic, endocrine, hematopoietic (any kind of anemia), asthma, mental or organic disease. Those suffering from muscular trauma 21 days before the beginning of the study.
* Requirement of any kind of medication during the course of the study, except study medication.
* History of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer.
* Exposure to medications known as inducers or inhibitors of hepatic enzymes or administration of potentially toxic medication in the 30 days before the study beginning.
* Administration of any medication in the 14 days or 5 half-lives (whatever longer) previous to the beginning of the study.
* Hospitalization for any cause in the seven months before the beginning of the study.
* Administration of investigational drugs in the 60 days before the study.
* Allergy to any medication, food, or substance.
* Alcohol ingestion or intake of beverages containing xanthines (coffee, tea, cocoa, chocolate, mate, cola drinks) or ingestion of charcoal grilled food or grapefruit or orange juice in the 72 hours before the hospitalization or tobacco smoking in the 72 hours before the beginning of the study.
* Blood donation or loss => 450 ml in the 60 days before the beginning of the study.
* History of drug or alcohol abuse.
* Special diet requirement, for instance vegetarian diet.
* Inability to understand nature, aims, and possible consequences of the study.
* Non-cooperative attitude during the study.
* Positive anti-doping or pregnancy test.
* Breast-feeding.
* Females on hormonal treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2010-12-10 (Actual); Study Completion 2010-12-10 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of alprazolam | 0.0, 0.167, 0.333, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 9.0, 12.0, 18.0, 22.0, 36.0, 48.0, 60.0, and 72.0 hours postdosage
  Pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of alprazolam | 0.0, 0.167, 0.333, 0.5, 0.75, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 9.0, 12.0, 18.0, 22.0, 36.0, 48.0, 60.0, and 72.0 hours postdosage
  Pharmacokinetcis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 116937 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116937?search=study&search_terms=116937#rs